CLINICAL TRIAL: NCT06998927
Title: Proportional Assist Ventilation Plus and Estimation of Respiratory Effort in Critically Ill Patients During the Transition to Spontaneous Ventilation: A Prospective Cohort Study
Brief Title: Proportional Assist Ventilation Plus and Estimation of Respiratory Effort During the Transition to Spontaneous Ventilation
Acronym: PAV+ and WOB
Status: Active, not recruiting | Type: Observational
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Gustavo Plotnikow, Head of Physical and Respiratory Care Department, ICU, Argentinian Intensive Care Society
Other Study IDs: CRIHB 12048
Record Dates: First submitted 2025-05-21; First posted 2025-05-31 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Effort; Proportional Assist Ventilation; Work of Breathing
MeSH Terms: interventions — EAP protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically ill patients during the transition from controlled mechanical ventilation to spontaneous
  Interventions: Other: Application of Proportional Assist Ventilation Plus (PAV+) at three support levels (20%, 50%, 70%) to assess ventilator-displayed work of breathing and its correlation with physiologic measures.

INTERVENTIONS:
Other: Application of Proportional Assist Ventilation Plus (PAV+) at three support levels (20%, 50%, 70%) to assess ventilator-displayed work of breathing and its correlation with physiologic measures. — This intervention is distinguished by applying Proportional Assist Ventilation Plus (PAV+) at three support levels (20%, 50%, 70%) within the same patient, allowing a stepwise analysis of its effect on work of breathing. It uses real-time ventilator-displayed work of breathing, a noninvasive and underexplored tool, correlated with multiple physiological parameters such as esophageal pressure, Pocc, and P0.1. This within-subject design controls for interindividual variability, improving the precision of the analysis. Focusing on patients with spontaneous respiratory effort facilitates clinical application to optimize personalized ventilatory support. Thus, the study provides novel data to adjust support levels according to the patient's actual effort and to validate ventilator measurements against reference physiological indicators.

SUMMARY:
In intensive care units, many critically ill patients need help from a machine called a ventilator to breathe. Once these patients start to recover, doctors try to gradually reduce this support and help them breathe on their own again. However, not all patients are ready to be taken off the ventilator right away. During this transition, it's important to find the right amount of help-enough to support their breathing, but not so much that the machine does all the work for them.

This study focuses on a special type of ventilator setting called Proportional Assist Ventilation Plus (PAV+). Unlike traditional modes, which give a fixed level of support, PAV+ adjusts the amount of help it gives based on how hard the patient is trying to breathe. The more effort a patient makes, the more support the machine provides-and vice versa. This can make breathing feel more natural and may protect the lungs and breathing muscles during recovery.

Modern ventilators also display a measurement called "Work of Breathing," which tells how much effort the patient is using to breathe. This study wants to find out whether this measurement from the ventilator is a reliable way to monitor a patient's breathing effort, compared to other more invasive or complex methods.

The research will include 20 adult patients who are recovering in the ICU and have been on mechanical ventilation for more than 48 hours. All patients will have already met some criteria showing they're ready to begin breathing more on their own, but are not quite ready to have the breathing tube removed.

Each patient will go through different levels of PAV+ support, and researchers will record how much effort they make to breathe using several methods, including special pressure sensors and data from the ventilator.

The goal of the study is to better understand how to measure breathing effort safely and easily, and to improve how we support patients as they recover the ability to breathe on their own. If successful, this could help reduce complications and improve recovery for people on ventilators.

There are no added risks or costs for the patients involved. All equipment used in the study is already part of regular ICU care. Participation requires informed consent and the privacy of all participants will be fully protected.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 yrs) requiring invasive MV >48 hrs
* Meeting spontaneous breathing transition criteria:

  * Hemodynamic stability (NE <0.1 μg/kg/min)
  * Spontaneous breathing efforts
  * RASS -2 to +1
  * FiO₂ <50% or PaO₂ >60mmHg with PEEP ≤10cmH₂O
* Pre-existing esophageal balloon
* Tolerates spontaneous modes >5 mins
* Signed informed consent

Exclusion Criteria:

* Meets extubation criteria
* Hemodynamic instability
* Psychomotor agitation (RASS >+1)
* Bronchopleural fistula
* Severe weakness (MRC <36)
* Neuromuscular disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This prospective cohort study will enroll critically ill adults (>18years) requiring prolonged mechanical ventilation (>48 hours) at Hospital Británico de Buenos Aires' ICU. Participants represent a diverse urban population with complex respiratory failures (post-operative, pneumonia, ARDS, COPD or chronic cardiopulmonary exacerbations) transitioning to spontaneous breathing. The ICU, staffed by PAV+-trained specialists and equipped with Puritan Bennett™ ventilators/FluxMed® monitoring, provides a representative Latin American setting for studying challenging weaning cases.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Ventilator-Measured Work of Breathing Tool and and invasive respiratory effort markers | From enrollment to the end of measurents at 3 hours
  Correlation between non-invasive WOB (measured by Puritan Bennett™ ventilators tool) and invasive metrics (Pes/PTPes via esophageal catheter, in cmH₂O and cmH₂O·s) during PAV+. Analyzed across 3 assistance levels (20%/50%/70%) to validate ventilator-based effort monitoring.

SECONDARY OUTCOMES:
Pocc (expiratory occlusion pressure in cmH₂O) during PAV+ analyzed across 3 assistance levels (20%/50%/70%) to validate ventilator-based effort monitoring. | From enrollment to the end of measurements at 3 hours
  Validate ventilator-measured WOB against Pocc (cmH₂O) in PAV+ measures compared at 20%/50%/70% assistance to assess non-invasive monitoring accuracy.
P0.1 (inspiratory occlusion pressure at 100 mseg in cmH₂O) during PAV+ analyzed across 3 assistance levels (20%/50%/70%) to validate ventilator-based effort monitoring. | From enrollment to the end of measurements at 3 hours
  Validate ventilator-measured WOB against P0.1 (cmH₂O) in PAV+ measures compared at 20%/50%/70% assistance to assess non-invasive monitoring accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Británico de Buenos Aires, CABA, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arellano DH, Brito R, Morais CCA, Ruiz-Rudolph P, Gajardo AIJ, Guinez DV, Lazo MT, Ramirez I, Rojas VA, Cerda MA, Medel JN, Illanes V, Estuardo NR, Bruhn AR, Brochard LJ, Amato MBP, Cornejo RA. Pendelluft in hypoxemic patients resuming spontaneous breathing: proportional modes versus pressure support ventilation. Ann Intensive Care. 2023 Dec 20;13(1):131. doi: 10.1186/s13613-023-01230-w. PMID 38117367
- [Background] Spinazzola G, Ferrone G, Costa R, Festa O, Piastra M, Bello G, Amato MF, Rossi M, Conti G. "Evaluation of Different Inspiratory Efforts in a Pediatric Model of Healthy Lung and Pediatric Acute Respiratory Distress Syndrome During Optimized Pressure Support Ventilation and Proportional Assist Ventilation Plus (PAV+): A Bench Study. Pediatr Pulmonol. 2025 Mar;60(3):e71027. doi: 10.1002/ppul.71027. PMID 40042134
- [Background] Gerson EAM, Dominelli PB, Leahy MG, Kipp S, Guenette JA, Archiza B, Sheel AW. The effect of proportional assist ventilation on the electrical activity of the human diaphragm during exercise. Exp Physiol. 2023 Feb;108(2):296-306. doi: 10.1113/EP090808. Epub 2022 Nov 24. PMID 36420595
- [Background] Fazio SA, Lin G, Cortes-Puch I, Stocking JC, Tokeshi B, Kuhn BT, Adams JY, Harper R. Work of Breathing During Proportional Assist Ventilation as a Predictor of Extubation Failure. Respir Care. 2023 Aug;68(8):1049-1057. doi: 10.4187/respcare.10225. Epub 2023 May 9. PMID 37160340
- [Background] Amargiannitakis V, Gialamas I, Pediaditis E, Soundoulounaki S, Prinianakis G, Vaporidi K, Akoumianaki E, Proklou A, Alexopoulou C, Georgopoulos D, Kondili E. Validation of a Proposed Algorithm for Assistance Titration During Proportional Assist Ventilation With Load-Adjustable Gain Factors. Respir Care. 2020 Jan;65(1):36-44. doi: 10.4187/respcare.06988. Epub 2019 Sep 17. PMID 31530626
- [Background] Bertoni M, Telias I, Urner M, Long M, Del Sorbo L, Fan E, Sinderby C, Beck J, Liu L, Qiu H, Wong J, Slutsky AS, Ferguson ND, Brochard LJ, Goligher EC. A novel non-invasive method to detect excessively high respiratory effort and dynamic transpulmonary driving pressure during mechanical ventilation. Crit Care. 2019 Nov 6;23(1):346. doi: 10.1186/s13054-019-2617-0. PMID 31694692
- [Background] de Vries HJ, Tuinman PR, Jonkman AH, Liu L, Qiu H, Girbes ARJ, Zhang Y, de Man AME, de Grooth HJ, Heunks L. Performance of Noninvasive Airway Occlusion Maneuvers to Assess Lung Stress and Diaphragm Effort in Mechanically Ventilated Critically Ill Patients. Anesthesiology. 2023 Mar 1;138(3):274-288. doi: 10.1097/ALN.0000000000004467. PMID 36520507
- [Background] Sassoon CS, Light RW, Lodia R, Sieck GC, Mahutte CK. Pressure-time product during continuous positive airway pressure, pressure support ventilation, and T-piece during weaning from mechanical ventilation. Am Rev Respir Dis. 1991 Mar;143(3):469-75. doi: 10.1164/ajrccm/143.3.469. PMID 2001053
- [Background] Charlson ME, Charlson RE, Peterson JC, Marinopoulos SS, Briggs WM, Hollenberg JP. The Charlson comorbidity index is adapted to predict costs of chronic disease in primary care patients. J Clin Epidemiol. 2008 Dec;61(12):1234-1240. doi: 10.1016/j.jclinepi.2008.01.006. Epub 2008 Jul 10. PMID 18619805
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Baydur A, Behrakis PK, Zin WA, Jaeger M, Milic-Emili J. A simple method for assessing the validity of the esophageal balloon technique. Am Rev Respir Dis. 1982 Nov;126(5):788-91. doi: 10.1164/arrd.1982.126.5.788. PMID 7149443
- [Background] Hermans G, Clerckx B, Vanhullebusch T, Segers J, Vanpee G, Robbeets C, Casaer MP, Wouters P, Gosselink R, Van Den Berghe G. Interobserver agreement of Medical Research Council sum-score and handgrip strength in the intensive care unit. Muscle Nerve. 2012 Jan;45(1):18-25. doi: 10.1002/mus.22219. PMID 22190301
- [Background] Beloncle F, Akoumianaki E, Rittayamai N, Lyazidi A, Brochard L. Accuracy of delivered airway pressure and work of breathing estimation during proportional assist ventilation: a bench study. Ann Intensive Care. 2016 Dec;6(1):30. doi: 10.1186/s13613-016-0131-y. Epub 2016 Apr 14. PMID 27076185
- [Background] Vaporidi K, Psarologakis C, Proklou A, Pediaditis E, Akoumianaki E, Koutsiana E, Chytas A, Chouvarda I, Kondili E, Georgopoulos D. Driving pressure during proportional assist ventilation: an observational study. Ann Intensive Care. 2019 Jan 3;9(1):1. doi: 10.1186/s13613-018-0477-4. PMID 30603960
- [Background] Akoumianaki E, Prinianakis G, Kondili E, Malliotakis P, Georgopoulos D. Physiologic comparison of neurally adjusted ventilator assist, proportional assist and pressure support ventilation in critically ill patients. Respir Physiol Neurobiol. 2014 Nov 1;203:82-9. doi: 10.1016/j.resp.2014.08.012. Epub 2014 Aug 26. PMID 25169117
- [Background] Schmidt M, Kindler F, Cecchini J, Poitou T, Morawiec E, Persichini R, Similowski T, Demoule A. Neurally adjusted ventilatory assist and proportional assist ventilation both improve patient-ventilator interaction. Crit Care. 2015 Feb 25;19(1):56. doi: 10.1186/s13054-015-0763-6. PMID 25879592
- [Background] Doorduin J, Sinderby CA, Beck J, van der Hoeven JG, Heunks LM. Assisted Ventilation in Patients with Acute Respiratory Distress Syndrome: Lung-distending Pressure and Patient-Ventilator Interaction. Anesthesiology. 2015 Jul;123(1):181-90. doi: 10.1097/ALN.0000000000000694. PMID 25955983
- [Background] Suarez-Sipmann F; Acute Respiratory Failure Working Group of the SEMICYUC. New modes of assisted mechanical ventilation. Med Intensiva. 2014 May;38(4):249-60. doi: 10.1016/j.medin.2013.10.008. Epub 2014 Feb 5. English, Spanish. PMID 24507472
- [Background] Jubran A, Van de Graaff WB, Tobin MJ. Variability of patient-ventilator interaction with pressure support ventilation in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1995 Jul;152(1):129-36. doi: 10.1164/ajrccm.152.1.7599811.
- [Background] Dianti J, Fard S, Wong J, Chan TCY, Del Sorbo L, Fan E, Amato MBP, Granton J, Burry L, Reid WD, Zhang B, Ratano D, Keshavjee S, Slutsky AS, Brochard LJ, Ferguson ND, Goligher EC. Strategies for lung- and diaphragm-protective ventilation in acute hypoxemic respiratory failure: a physiological trial. Crit Care. 2022 Aug 29;26(1):259. doi: 10.1186/s13054-022-04123-9. PMID 36038890
- [Background] Xirouhaki N, Kondili E, Mitrouska I, Siafakas N, Georgopoulos D. Response of respiratory motor output to varying pressure in mechanically ventilated patients. Eur Respir J. 1999 Sep;14(3):508-16. doi: 10.1034/j.1399-3003.1999.14c06.x. PMID 10543268
- [Background] Alberti A, Gallo F, Fongaro A, Valenti S, Rossi A. P0.1 is a useful parameter in setting the level of pressure support ventilation. Intensive Care Med. 1995 Jul;21(7):547-53. doi: 10.1007/BF01700158. PMID 7593895
- [Background] Kataoka J, Kuriyama A, Norisue Y, Fujitani S. Proportional modes versus pressure support ventilation: a systematic review and meta-analysis. Ann Intensive Care. 2018 Dec 10;8(1):123. doi: 10.1186/s13613-018-0470-y. PMID 30535648
- [Background] MacIntyre NR. Respiratory function during pressure support ventilation. Chest. 1986 May;89(5):677-83. doi: 10.1378/chest.89.5.677. PMID 3698697
- [Background] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Background] Plotnikow GA, Gogniat E, Accoce M, Navarro E, Dorado JH; EpVAr study group. Epidemiology of mechanical ventilation in Argentina. The EpVAr multicenter observational study. Med Intensiva (Engl Ed). 2022 Jul;46(7):372-382. doi: 10.1016/j.medine.2022.05.002. Epub 2022 May 31. PMID 35660286
- [Background] Esteban A, Anzueto A, Alia I, Gordo F, Apezteguia C, Palizas F, Cide D, Goldwaser R, Soto L, Bugedo G, Rodrigo C, Pimentel J, Raimondi G, Tobin MJ. How is mechanical ventilation employed in the intensive care unit? An international utilization review. Am J Respir Crit Care Med. 2000 May;161(5):1450-8. doi: 10.1164/ajrccm.161.5.9902018. PMID 10806138
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Perez J, Accoce M, Dorado JH, Gilgado DI, Navarro E, Cardoso GP, Telias I, Rodriguez PO, Brochard L. Failure of First Transition to Pressure Support Ventilation After Spontaneous Awakening Trials in Hypoxemic Respiratory Failure: Influence of COVID-19. Crit Care Explor. 2023 Aug 25;5(9):e0968. doi: 10.1097/CCE.0000000000000968. eCollection 2023 Sep. PMID 37644972
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684